CLINICAL TRIAL: NCT01455662
Title: Relationship Between Lactate and Venous Oxygen Saturation Gradient of Carbon Dioxide in Patients With Post Cardio Respiratory Syndrome
Brief Title: Relationship Between Tissue Markes in Patients With Post Cardio Respiratory Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Vanessa Martins de oliveira, Principal Investigator, Hospital Nossa Senhora da Conceicao
Other Study IDs: 10086
Record Dates: First submitted 2011-09-28; First posted 2011-10-20 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- all patients after cardiac arrest

SUMMARY:
There is a correlation between hospital mortality and changes in markers of tissue perfusion, lactate, and venous oxygen saturation and carbon dioxide gradient.

DETAILED DESCRIPTION:
Evaluation of the serum carbon dioxide gradient (GapCO2), central venous saturation (ScvO2) and the clearance of serum lactate (Clac) in predicting hospital mortality after cardiac arrest syndrome (post-PCR).

Prospective study, unicenter - Intensive Care Unit - HNSC. Period: May/2010 to June/2011. Serial assessment of GapCO2 of ScvO2 Clac and the first 72 hours post-PCR. Excluded under 18, survival of less than 6HS, pregnant women, traumatized, post-operative hypothermia and liver disease. T-student test, 95% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the intensive care unit after cardiopulmonary arrest with any pace

Exclusion Criteria:

pregnant women, traumatized, post-operative(less 7 days), hypothermia and liver disease.

* patients hospitalized in the intensive care unit with more than 6 hours post cardiac arrest
* less 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in the intensive care unit after cardiopulmonary arrest
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 year

SECONDARY OUTCOMES:
correlation of clearance markers of perfusion with the use of vasopressor and positive fluid balance | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Oliveira, MD, Principal Investigator — Conceição Hospital; Diego F Riveiro, MD, Principal Investigator — Hospital Nossa Senhora da Conceição
Locations (1):
- Conceição Hospital, Porto Alegre, Rio Grande do Sul, Brazil